CLINICAL TRIAL: NCT07088510
Title: A Randomized Control Trial Investigating Hysteroscopic Resection Versus Manual Vacuum Aspiration for Early Pregnancy
Brief Title: Hysteroscopic Resection Versus Manual Vacuum Aspiration for Early Pregnancy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Joseph Findley MD, Assistant Professor, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY20240983
Record Dates: First submitted 2025-07-19; First posted 2025-07-28 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Miscarriage in First Trimester
Keywords: hysteroscopy; dilation and curettage; Manual Vacuum Aspiration
MeSH Terms: conditions — Dilatation, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hysteroscopy (Experimental): Participants will undergo hysteroscopic resection of early pregnancy loss under monitored anesthesia care.
  Interventions: Procedure: Hysteroscopic resection
- Manual Vacuum Aspiration (Active Comparator): Participants will undergo manual vacuum aspiration of early pregnancy loss under monitored anesthesia care.
  Interventions: Procedure: Manual Vacuum Aspiration

INTERVENTIONS:
Procedure: Hysteroscopic resection — Participants will undergo a hysteroscopy where a camera is placed on the inside of the uterus. Then a resector will be used to remove the pregnancy loss under direct visualization.
  Arms: Hysteroscopy
Procedure: Manual Vacuum Aspiration — Participants will undergo a manual vacuum aspiration with ultrasound guidance for treatment of early pregnancy loss. This is when pregnancy loss is suctioned by a machine from the uterus.
  Arms: Manual Vacuum Aspiration

SUMMARY:
Early pregnancy loss happens when a pregnancy that is not developing properly is found on an ultrasound before 12 weeks and 6 days. This type of loss occurs in about 10% of pregnancies. There are three main ways to treat this: waiting for it to pass naturally, using medication, or having surgery. Surgery is the most effective, working 99% of the time, compared to waiting (80% effective in 8 weeks) and medication (71-84% effective). Currently, surgery involves dilation of the cervix and curettage (removal of pregnancy tissue) with suction provided either from a manual hand-held pump or a machine. For the purposes of this study, a manual vacuum aspirator (or hand-held pump) will be used with ultrasound guidance.

There is also another method called hysteroscopic resection, where the doctor uses a special camera to directly see and remove any pregnancy tissue from your uterus. Patients often want the quickest way to resolve the pregnancy loss, and physicians are unsure which surgical method is the best. It's also unclear if one type of surgery causes less scar tissue inside the uterus, affects the ability to test the tissue for genetic issues, or impacts how soon a patient can start fertility treatments again.

This study aims to find out if hysteroscopic resection provides faster resolution and creates less scar tissue compared to the manual vacuum aspiration.

DETAILED DESCRIPTION:
Early pregnancy loss is when a nonviable intrauterine pregnancy is diagnosed on ultrasound prior to 12 weeks and 6 days of gestation and occurs in 10% of pregnancies. There are typically three treatment modalities: expectant management, medical management, or surgical management. Surgical management is 99% effective in comparison to expectant management (80% resolution within 8 weeks) and medical management (71-84%). Current standard surgical management includes manual vacuum aspiration or suction dilation and curettage with or without ultrasound guidance. Hysteroscopic resection of retained products of conception (RPOC) has been studied. A recent randomized control trial comparing this to vacuum curettage showed hysteroscopic resection of RPOC had an increase in completeness of removal of the RPOC and decreased need for additional treatment with either a second hysteroscopy or vacuum curettage. Although detailed in 1 case report and performed nationally, hysteroscopic resection in comparison to manual vacuum aspiration of early pregnancy loss has not been investigated. Potential benefits of hysteroscopic resection in comparison to manual vacuum aspiration include faster return to negative bHCG, decreased risk of intrauterine adhesion formation post-operatively, and decreased risk of retained products of conception. Furthermore, 50% of early pregnancy losses are due to fetal chromosomal abnormalities. Thus, diagnosis of a chromosomal abnormality can both provide information for the patient and allow for guidance of pregnancy treatment in the future. A retrospective chart review determined that obtaining fetal genetics is less likely to be contaminated with maternal tissue and is more likely to detect fetal chromosomes when the products of conception were biopsied hysteroscopically prior to suction dilation and curettage rather than when the pregnancy is terminated solely with suction dilation and curettage. Thus, hysteroscopic resection of early pregnancy loss may provide cytogenetic information that may not be obtained with a manual vacuum aspiration (similar technique as suction dilation and curettage, using manual suction instead of electric suction). This study aims to find out if hysteroscopic resection provides faster resolution of the pregnancy loss, creates less scar tissue, and improves genetic testing in comparison to manual vacuum aspiration.

ELIGIBILITY:
Inclusion Criteria:

* Adult women age 18-55
* Ultrasound Diagnosis of Early Pregnancy Loss
* < 9 weeks gestational age as determined by ultrasound
* Singleton non-viable pregnancy
* Stated and willingness to comply with all study procedures and availability for the duration of the study
* Provision of signed and dated informed consent form
* Chose a surgical method of management for fetal loss

Exclusion Criteria:

* Pregnancy of Unknown Location
* Current, viable pregnancy
* Prior medical treatment for this early pregnancy loss
* Contraindications to surgical management
* Active infection (i.e. fever, chills, fundal tenderness)
* Pre-existing coagulopathies

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in beta human chorionic gonadotropin (bHCG) levels as measured by blood test | Baseline, 1 week post operation, 2 week post operation, 3 week post operation, 4 week post operation, 5 week post operation

SECONDARY OUTCOMES:
Number of uterine adhesions detected by follow up hysteroscopy | 4 weeks post operation
Number of post operative bleeding incidences as measured by nurse observation | Up to 1 hour post operation
Time in minutes to complete procedure | Up to 30 minutes
Number of retained products of conception as seen on follow up hysteroscopy | 1 month post operation
Number of additional treatments needed as measured by follow up hysteroscopy | 1 month post operation
Time in months to next fertility treatment | Up to 12 months
Number of completed cytogenetic results as measured genetic testing | Up to 1 month post operation

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Findley, MD, Principal Investigator — University Hospitals; Archana Ayyar, MD, Principal Investigator — University Hospitals
Locations (1):
- University Hospitals, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No